CLINICAL TRIAL: NCT03978611
Title: A Phase 1/2a Study to Evaluate the Safety, Tolerability, and Efficacy of Relatlimab Administered in Combination With Ipilimumab or Ipilimumab Alone in Participants With Unresectable or Metastatic Melanoma Who Have Progressed on Anti-PD-1 Therapy
Brief Title: A Study to Assess Safety of Relatlimab With Ipilimumab in Participants With Advanced Melanoma Who Progressed on Anti-Programmed Cell Death Protein 1 (Anti-PD-1) Treatment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA224-083; 2019-000132-25 (EudraCT Number)
Expanded Access: NCT05170659 (No longer available)
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — relatlimab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1: Dose Escalation Phase (Experimental)
  Interventions: Drug: Relatlimab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Relatlimab — Specified dose on specified days
  Other Names: BMS-986016
Drug: Ipilimumab — Specified dose on specified days

SUMMARY:
The primary purpose of this study is to characterize the safety, tolerability, and dose-limiting toxicities (DLTs) of relatlimab in combination with ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

* Must have documented progression while on a prior anti-programmed cell death protein 1 (PD-1) containing regimen limited to Nivolumab or Pembrolizumab
* Must have histologically confirmed advanced unresectable (Stage III) or metastatic (Stage IV) melanoma, as per (AJCC) staging system
* Tumor tissue from an unresectable or metastatic site of disease must be provided for biomarker analyses
* Eastern Cooperative Oncology Group (ECOG) 0-1

Exclusion Criteria:

* History of uveal melanoma
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome
* Prior treatment with ipilimumab, relatlimab, or any other cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) or lymphocyte-activation gene 3 (LAG-3) targeted agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Follow-up Period (100 days after 34 cycles [1 cycle is of 3 weeks])
Number of Participants with Serious Adverse Events (SAEs) | Up to Follow-up Period (100 days after 34 cycles [1 cycle is of 3 weeks])
Number of Participants With Adverse Events Including Dose Limiting Toxicity | Up to 28 days after last study drug dose (approximately up to 2 years)
Number of Participants with AEs resulting in Discontinuation | Up to end of study (approximately 2.4 years)
Number of Participants with AEs resulting in Death | Up to end of study (approximately 2.4 years)
Number of Participants with AEs resulting in Laboratory Abnormalities | Up to end of study (approximately 2.4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (28):
- United States (8):
  - Local Institution - 0023, Tucson, Arizona
  - Local Institution - 0002, Los Angeles, California
  - Local Institution - 0005, Los Angeles, California
  - Local Institution - 0001, Santa Monica, California
  - Local Institution - 0015, Miami, Florida
  - Local Institution - 0004, Chicago, Illinois
  - Local Institution - 0003, Ann Arbor, Michigan
  - Local Institution - 0008, Morristown, New Jersey
- Belgium (4):
  - Local Institution - 0018, Brussels, Brussels Capital
  - Local Institution - 0017, Antwerp
  - Local Institution - 0016, Brussels
  - Local Institution - 0038, Brussels
- Local Institution - 0044, Ottawa, Ontario, Canada
- Germany (7):
  - Local Institution - 0037, Erlangen
  - Local Institution - 0034, Essen
  - Local Institution - 0036, Gera
  - Local Institution - 0035, Hanover
  - Local Institution - 0033, Heidelberg
  - Local Institution - 0032, Lübeck
  - Local Institution - 0040, Nuremberg
- Italy (2):
  - Local Institution - 0053, Padua
  - Local Institution - 0055, Siena
- Spain (6):
  - Local Institution - 0026, Barcelona
  - Local Institution - 0030, Córdoba
  - Local Institution - 0031, Donostia / San Sebastian
  - Local Institution - 0027, Hospitalet de Llobregat - Barcelona
  - Local Institution - 0029, Madrid
  - Local Institution - 0028, Valencia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com